Renata Medical Version C PTC-0009 07-November-2022





## GROWTH: A Multicenter Pivotal Study of Neonatal, Infant, and Young Child Vascular Stenoses Studying the Renata Minima Stent

## **Clinical Protocol**

**Protocol Number: PTC-0009** 

NCT Number: NCT05086016

Version C

11/07/2022

Study Sponsor: Renata Medical

**Proprietary - Uncontrolled if Printed** 

## **Protocol Synopsis**

| <b>Protocol Number</b> | PTC-0009 |
|---|---|
| Title | Multicenter Pivotal Study of Neonate, Infant, and Young Child<br>Vascular Stenoses Studying the Renata Minima Stent |
| Phase | Pivotal Study |
| Sponsor | Renata Medical |
| <b>Investigational Device</b> | Minima Stent |
| Study Objectives | To assess device performance and clinical safety and effectiveness of the Minima Stent in neonates, infants and young children requiring intervention for coarctation of the aorta or pulmonary artery stenosis who are indicated for treatment. |
| Study Design | Single arm, prospective, non-randomized, multi-center, open-label, Pivotal study. |
| Study Population | The study population will be comprised of patients with a clinically relevant pulmonary artery or aortic vascular stenosis who are indicated for treatment. For each treatment location (pulmonary artery or aortic vascular), a minimum of 10 patients will be treated. |
| Inclusion<br>Criteria | <ul> <li>Inclusion criteria include: <ul> <li>The subject's legally authorized representative has been informed of the nature of the clinical investigation, agrees to its provisions, and has provided written informed consent</li> <li>Requiring treatment* of:</li></ul></li></ul> |
| Exclusion Criteria | Exclusion criteria include: |
| | • Active bloodstream infection requiring antibiotic therapy within 3 days prior to stent implantation |

| | History of or active endocarditis (active treatment with antibiotics) within 180 days prior to stent implantation |
|---|---|
| | Aortic or pulmonary artery aneurysm in the location targeted for treatment |
| | Body weight < 1.5 kg |
| | Anatomic location of lesion judged by the investigator to not lend to the safe placement of a stent |
| | Target vessels larger or smaller than the Minima System balloon size ranges |
| | Known genetic syndrome known to be associated with vasculopathies such as but not limited to Williams syndrome, Loeys-Dietz syndrome, etc |
| | Clinical scenario requiring that more than one vessel needs stent implantation at the time of the trial procedure. |
| | Currently participating in an investigational drug study or another device study |
| | Major or progressive non-cardiac disease resulting in a life expectancy of less than six months |
| | Known hypersensitivity to aspirin or heparin and cannot be treated with other antiplatelet and/or antithrombotic medications |
| | Known hypersensitivity to cobalt-chromium or contrast media that cannot be adequately pre-medicated |
| Number of Subjects | Maximum of 42 US subjects |
| Number of Study Sites | 8 US sites, with the possibility of additional Japanese and/or European Union sites pending the appropriate regulatory approvals. |
| <b>Location of Study Sites</b> | Children's Hospital Los Angeles |
| | Cedars Sinai Medical Center |
| | Seattle Children's Hospital |
| | Cincinnati Children's Hospital |
| | Boston Children's Hospital |
| | Nationwide Children's Hospital |
| | Le Bonheur Children's Hospital |
| Visit Schedule | Screening/baseline, discharge, 1 month, 3 months, 6 months, 12 months, and annually thereafter through 5 years |

| | Enrollment is expected to take up to 6 months and will be ongoing throughout the study. |
|---|---|
| Primary Efficacy Endpoint | <ul> <li>The primary efficacy endpoint will be assessed as the rate of clinical success, with the performance goal defined as a clinical success rate of greater than 77%.</li> <li>Clinical success is defined as: <ul> <li>Stenosis relief, defined by stent outer diameter ≥ 75% of the surrounding vessel immediately after deployment.</li> <li>Freedom from open surgical intervention required to treat Minima Stent disfunction through 6 months.</li> <li>Maintenance of stented vessel diameter ≥ 50% of post-implant diameter at 6 months; as measured using CT angiography and/or angiography.</li> </ul> </li> </ul> |
| Primary Safety Endpoint | The primary safety endpoint will be assessed as the percentage of cases with freedom from procedure- or device-related SAEs resulting in an event listed below, with the performance goal defined as greater than 78% of cases: O Death O Cardiac arrest and/or emergency ECMO cannulation O Stroke O Limb loss O Vessel dissection of target lesion O Device thrombosis/occlusion O Cardiac perforation requiring percutaneous or open surgical intervention O Persistent cardiac arrhythmia requiring a pacemaker |
| Secondary Efficacy<br>Endpoints | <ul> <li>Peak-to-peak pressure gradient (ventricle to arterial or arterial to arterial) &lt; 20 mmHg after stent placement, when applicable.</li> <li>Successful stent re-dilation (when indicated) at recatheterization, defined as an increase in the intra stent angiographic luminal diameter within 2mm of the adjacent native vessel diameter immediately after re-dilation.</li> </ul> |
| Secondary Safety Endpoints | <ul> <li>Freedom from stent embolization or migration through 6 months.</li> <li>Freedom from stent fracture that led to reintervention through 6 months</li> <li>Freedom from non-elective Minima Stent explant at 90-days post re-dilation</li> <li>Freedom from procedure- or device-related SAE during redilation that results in the following: <ul> <li>Death</li> <li>Cardiac arrest and/or emergency ECMO cannulation</li> <li>Stroke</li> <li>Limb loss</li> <li>Vessel dissection of target lesion</li> </ul> </li> </ul> |

| | <ul> <li>Device thrombosis/occlusion</li> <li>Cardiac perforation requiring percutaneous or open surgical intervention</li> <li>Persistent cardiac arrhythmia requiring a pacemaker</li> </ul> |
|---|---|
| Sample Size Considerations | The study intends to enroll a maximum of 42 subjects within the United States. For each treatment location (pulmonary artery or aortic vascular), a minimum of 10 patients will be treated. Additionally, no site will be permitted to enroll more than one third of the total subjects implanted in the study. The chosen sample size is appropriate, as it allows for the analysis of each co-primary endpoint, with the appropriate power level. See |
| Statistical Analysis Methods | Descriptive statistics will be the primary analysis method. The proportion of subjects with device success will be calculated along with the associated 95% confidence interval. Other categorical endpoints will be described with percentages. Continuous variables will be presented as mean with the standard deviation or median. Time-to-event endpoints will be described with Kaplan Meier graphs as appropriate. Other statistical analysis methods and graphing methods can be used in addition to those listed above, as appropriate. |